CLINICAL TRIAL: NCT06522529
Title: SUMAMOS EXCELENCIA Project: Assessment of Implementation of Best Practices in a National Health System (Thrid Edition)
Brief Title: Sumamos Excelencia Project: Implementation of Best Practices in Clinical Practice (Thrid Edition)
Acronym: SE24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: The Spanish Centre for Evidence Based Nursing and Healthcare (Unknown)
Responsible Party: Principal Investigator, Teresa Moreno Casbas, Doctor, Instituto de Salud Carlos III
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SE_CECBE_2024
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Pain; Obesity, Childhood; Breast Feeding; Incontinence, Urinary; Smoking Cessation; Pressure Injury; Fall
Keywords: Implementation; Implementation science; Evidence-based practice; Nursing; Quality of Health Care
MeSH Terms: conditions — Pain; Pediatric Obesity; Breast Feeding; Urinary Incontinence; Smoking Cessation; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, uncontrolled, before-and-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Quasi-experimental uncontrolled, before-and-after. (Experimental): The intervention will consist of the use of a multifaceted implementation strategy based in the continuous quality improvement cycle model and in implementation science theories, model and frameworks to be developed in clinical practice according to the study unit in question and the scope of action.
  Interventions: Other: Multifaceted implementation strategy

INTERVENTIONS:
Other: Multifaceted implementation strategy — The multifaceted implementation strategy consist in a process of improvement by reference to a prior baseline clinical audit. It implies a local context analysis, identifying barriers to improvements in clinical practice, and developing and implementing a plan of action for improving adherence to pre-established criteria. The goal is to establish interprofessional processes within the teams, in order to: examine the barriers that hinder the use of evidence in fostering best practices; and contribute to the development of implementation programmes for overcoming such obstacles.

SUMMARY:
There is a gap between research and clinical practice, leading to variability in decision-making. Multifaceted implementation strategies are for improving implementation of best practices. Quasi-experimental, multicentre, before and after. Primary care, hospital units and nursing homes, and the patients attended at both. Implementation of evidence-based recommendations by application of a multifaceted implementation strategy (training, audit, context analysis, local strategies design, feedback, facilitation). Data will be collected at baseline and, during the first year of follow up, at months (4,8,12)

DETAILED DESCRIPTION:
Aim: To assess the effectiveness of implementing evidence-based recommendations using multifaceted implementation strategy on patient outcomes and healthcare quality. Design: Quasi-experimental, multicentre, before-and-after. Methods: NHS units and Nursing Homes, patients attended by them and professionals implementing the recommendations. Intervention: implementation of evidence-based recommendation with a multifaceted implementation strategy (training, audit, context analysis, local strategies design, feedback, facilitation). Variables: Process and outcome criteria with respect to assessment and management of pain, management of urinary incontinence, prevention of child obesity, promotion of breastfeeding, promotion of hand hygiene, smoking cessation intervention, pressure injury prevention, fall prevention, competencies in evidence-based practice, barriers to the implementation and strategies for overcoming them. Data will be collected at baseline and, during the first year of follow-up, at months 4, 8 and 12, with data on patients and indicators being drawn from clinical histories and records. Descriptive analysis and comparison of the effectiveness of the intervention by means of inferential analysis and analysis of trends across follow-up. 95% confidence level. This project is partially funded by The Spanish Centre for Evidence Based Nursing and Healthcare. Project duration 2024-2025.

This project is a third edition of The SUMAMOS EXCELENCIA Project: Assessment of Implementation of Best Practices in a National Health System (NCT05466656), with an improved design and new recommendation topics.

ELIGIBILITY:
Inclusion Criteria:

1. Unit inclusion criteria:

   * NHS units and nursing homes which voluntary adhere to the project.
   * NHS units and nursing homes providing direct patient care and commit to implement evidence-based recommendations on hand hygiene and one of the following topics: pain assessment and management, urinary incontinence management, obesity prevention and breastfeeding promotion, Smoking Cessation, falls prevention, pressure injuries prevention. For the purposes of this study, a "unit" is defined as any service, centre or institution that delivers health services to a homogeneous group of patients who share similar characteristics.
2. Patient inclusion criteria: The study will include all patients attended in the units participating in the study, who meet the following criteria, depending on the recommendations to be implemented in each unit:

   1. Pain:

      * People susceptible to suffering some type of pain regardless of age.
      * Patients treated in acute or chronic health institutions (Hospitals, Nursing Homes or Primary Care).
   2. Urinary incontinence:

      - Patients 18 years or older.

      - Patients with uncomplicated stress, urge or mixed urinary incontinence

      - At least 7 days of admission or possibility of continuity of care preferably up to 6 weeks.
   3. Obesity:

      * Babies and preschool children up to 12 years old.
      * For ages 2 to 12 years (inclusive), children must not be overweight or obese 1 year prior to baseline measurement (in February 2021 or at the closest review to February 2021 at which BMI is recorded).
      * Good general health.
   4. Breastfeeding:

      * Lactating people.
      * Healthy neonates of gestational age greater than 36 weeks, with birth weight greater than or equal to 2500 gr.
      * Couples and relatives within the support network.
      * Postpartum period and up to 6 months of life of the baby (183 days of life, included).
      * In primary care, only non-urgent care will be included.
   5. Smoking Cessation:

      - ≥ 18 years of age
      * Smokers
   6. Pressure injury prevention:

      - Adults population (≥ 18 years).
      * Admitted to hospitals, nursing homes or included in home care programmes.
      * Patients at risk of developing pressure injuries.
   7. Falls prevention:

      * Adults aged 65 years or older, and adults aged 18 years or older who may potentially present problems in walking as a result of neurological or traumatic diseases, medication, or who suffer from loss of strength or drowsiness.
   8. Hand hygiene:

      - All health professionals who care for patients in the units participating in the study.

      Exclusion Criteria:

      -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
ICU beds with alcohol-based preparations at the point of care | 15 months
  Availability of the alcohol-based preparations in the Intensive Care Units (Hospital care) as close as possible to the place where an activity that requires contact with the patient and/or their immediate environment is going to be carried out and without having to leave the patient's area. Point of care is the place where the patient, the health professional and the care or treatment that involves contact with the patient coincide. (Number of ICU beds in the unit, with base alcoholic preparations at the point of care / Number of ICU beds in the unit) x100
Hospital beds with alcohol-based preparations at the point of care | 15 months
  Availability of the alcohol-based preparations in the hospital units (excluding ICU beds) as close as possible to the place where an activity that requires contact with the patient and/or their immediate environment is going to be carried out and without having to leave the patient's area. Point of care is the place where the patient, the health professional and the care or treatment that involves contact with the patient coincide. (Number of hospitalization beds in the unit, with alcohol-based preparations at the point of care)/(Number of beds in the unit) x100
Consumption of alcohol-based preparations in Primary Care centers | 15 months
  Litres of alcohol-based preparations consumed in primary care centres. (Number of liters of alcohol-based preparations delivered in primary care / Total number of consultations in the evaluated period) x10000
Consumption of alcohol-based preparations in hospital units without admission | 15 months
  Litres of alcohol-based preparations consumed in hospital units without admission (outpatient consultations, day hospital, etc.). (Number of liters of alcohol-based preparations@delivered in a hospital unit without admission / Total number of consultations in the evaluated period) x1000
Consumption of alcohol-based preparations in Nursing Homes. | 15 months
  Litres of alcohol-based preparations consumed in Nursing Homes (Number of liters of alcohol-based preparations delivered in Nursing Homes / Total number of residents in the evaluated period) x100
Detection of pain at admission | 15 months
  Detection of pain at admission. (Total number of patients in whom pain detection was performed upon admission or at the start of care, and it is registered / Total number of patients discharged or attended in the collection period data) x100
Pain related to a procedure likely to cause pain | 15 months
  Detection of pain related to a procedure likely to cause pain. This indicator evaluates whether the assessment of pain linked to the painful procedure is carried out before and after the procedure, it is also recommended to assess pain during the procedure in cases where it is possible. (Total number of patients in whom pain has been detected after a procedure likely to cause pain, and is registered / Total number of patients in whom a procedure likely to cause pain has been performed in the data collection period data) x100
Pain after a change in the patient's clinical situation | 15 months
  Detection of pain after a change in the patient's clinical situation (clinical situation: significant clinical change, in the general condition of the patient or in their pain, which requires the referral of the patient to a professional with the skills to resolve it). (Total number of patients in whom pain has been detected after a change in their clinical situation, and it is registered / Total number of patients with a change in their clinical situation in the data collection period) x100
Pain intensity assessment | 15 months
  Pain assessment measured with a pain intensity assessment tool. (Total number of patients who have an assessment of pain intensity, and it is recorded / Total number of patients with positive detection of pain in the data collection period) x100
Comprehensive pain assessment | 15 months
  Comprehensive pain assessment takes into account various factors related to pain, including: location of pain, circumstances related to the onset of pain, type of pain, pain intensity, associated symptoms, effect of pain on activities, effect of pain on patient rest and sleep, treatment, relevant medical history, factors that influence pain management. To be considered a comprehensive assessment, at least 60% of the 10 criteria must be performed and recorded. (Total number of patients who have done a comprehensive pain assessment, and it is registered / Total number of patients with positive pain detection in the data collection period) x100
Pain management care plan | 15 months
  Establishing and implementing a pain management care plan for the patient based on the results of the person's assessment, which would include: pharmacological and non-pharmacological measures, the person's goals and appropriate and effective pain management strategies. (Total number of patients with a care plan for acute or chronic pain, and it is registered / Total number of patients with positive detection of pain or susceptible to have pain in the data collection period) x100
Patient or/and caregiver education on pain | 15 months
  Patient or/and caregiver education on the importance of communicating pain, pharmacological, physical and psychological pain management options, how to take the analgesic medication, manage the possible side effects and how the follow-up will be done and who can be consulted with possible doubts. (Total number of patients, family members or caregivers who have received education on pain management, at least once during the care process, and it is registered / Total number of patients with positive detection of pain or likely to have pain in the data collection period) x100
Intensity of pain on admission or in the first 24 hours after surgery or at the start of care | 15 months
  Intensity of pain on admission or in the first 24 hours after surgery or at the start of care measured in numerical format, with the value that corresponds to the scale used in the unit for the assessment of pain, units must indicate on the form the scale they have used. (Sum of pain intensity of patients with positive pain detection or likely to have pain / Total number of patients with assessed pain intensity in the data collection period)
Maximum pain | 15 months
  Maximum scored reported by patients and registered by nurses after pain intensity assessment using an assessment tool. Units must indicate on the form the assessment tool they have used. (Sum of the maximum intensity of pain during the stay or care of patients with positive detection of pain or likely to have pain / Total number of patients with pain intensity assessed in the data collection period)
Quantification assessment in active smokers | 15 months
  Quantitative assessment of the intensity of tobacco or tobacco products use measured with a validated tool (Total number of patients who have undergone a quantification assessment and it is recorded )/(Total number of patients with positive detection of active smoking @ in the period of data collection ) x100 Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
Comprehensive assessment of active smokers | 15 months
  Assessment carried out with a comprehensive and systematic approach, taking into account various factors related to smoking, such as: Motivation to quit smoking (measured with the Richmond test); Degree of nicotine dependence (measured with the full Fagerström test); Current nicotine withdrawal symptoms; Previous quit attempts; Current need for smoking cessation treatments; Factors influencing patient behaviour change. The criterion is met when at least 50% of the 6 criteria (at least 3) are fulfilled and recorded (Total number of patients who have had a comprehensive smoking assessment performed and recorded)/(Total number of patients with positive screening for active smoking in the data collection period )/(Total number of patients with a positive screening for active smoking in the data collection period ) x100
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
Comprehensive assessment of the non-active smoker | 15 months
  Assessment carried out with a comprehensive and systematic approach, taking into account various factors related to smoking, such as: Existence or not of current nicotine withdrawal symptoms; Relapses; Current stage of change; Other symptoms. The criterion is fulfilled when at least 3 of the 5 criteria are fulfilled and recorded (Total number of patients who have undergone a 'comprehensive non-active smoking assessment' and are recorded) / (Total number of non-active smoking patients in the data collection period) x100
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
Brief interventions performed | 15 months
  Number of brief interventions (BI) based on the 5 As and 5 Rs carried out in smoking patients. For a BI to be considered as having been carried out, the nurse must at least: convey the advice to 'stop smoking', advise the patient on smoking cessation, offer support and accompaniment and specific comments on the health risks related to smoking and the benefits related to smoking cessation. (Number of smoking patients who have undergone Brief Intervention)/(Total number of smoking patients seen in the data collection period) x100 Brief intervention (BI): Intervention in which there is a brief (less than five minutes) contact between the health care provider and the patient.
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
Derivation of the active smoking patient | 15 months
  Referral to smoking cessation follow-up consultations is considered to be referral to primary care consultations and/or specific monographic smoking cessation consultations. If the unit is capable of carrying out the follow-up, the recommendation will be considered to have been made when the follow-up is planned in the same unit (Number of smoking patients referred for smoking follow-up after being seen/(Total number of smoking patients seen in the period of data collection) x100
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
Expressed desire to quit smoking (active smokers) | 15 months
  Documented evidence of the patient's expressed desire to quit smoking after the brief intervention (Total number of patients who have expressed an expressed desire to quit smoking after the brief intervention)/(Total number of patients with positive smoking screening who have undergone a BI in the data collection period)/(Total number of patients with positive smoking screening who have undergone a BI in the data collection period)x100
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
  Brief intervention: Intervention in which there is a brief (less than five minutes) contact between the health care provider and the patient.
Maintenance of willingness to remain smoke-free (non-active smokers) | 15 months
  Documented evidence of the non-active smoker patient's expressed desire to maintain their willingness to remain smoke-free after the comprehensive assessment. (Total number of patients who maintain their willingness to quit smoking after comprehensive assessment of active smoking)/(Total number of non-active smoking patients who have undergone a comprehensive assessment in the data collection period)x100
  Active smoker: person who is currently smoking or has smoked in the last 30 days.
  Non-active smoker: smoked the last cigarette or similar product more than 30 days but less than 183 days (6 months) ago.
Pressure injuries risk assessment at the initiation of care | 15 months
  Assessment of the risk of pressure injuries in the first 24 hours of admission, after the initiation of care or the first visit in primary care with a structured, validated and reliable tool, together with clinical judgement (Total number of people with complete assessment of pressure injuries at admission or initiation of care)/(Total number of people with health care provision) x100.
Reassessment of the risk of pressure injuries | 15 months
  Reassessment of the risk of PBI: reassessment of the risk of developing pressure sores upon a significant clinical change in the person's general condition, change of caregiver, change of setting or care unit and at discharge; with a structured, validated and reliable tool, together with clinical judgement. (Total number of people with reassessment of pressure sores)/(Total number of people with health care provision) x100.
Nutritional screening of the person at risk of pressure injuries | 15 months
  Nutritional screening of the person at risk of developing pressure injuries with a structured, validated and reliable tool. (Total number of persons at risk of pressure injuries who have been nutritionally screened)/(Total number of persons at risk of pressure injuries) x100.
Support surfaces for the prevention of pressure injuries | 15 months
  Recording whether a support surface that meets the person's needs has been used to prevent the occurrence of pressure injuries (Total number of persons at risk of pressure injuries who have a support surface applied)/(Total number of persons at risk of pressure injuries) x100
Pressure injury prevention care plan | 15 months
  Establishing and implementing a pressure injury prevention care plan for the patient based on the results of the person's assessment, which would include: comprehensive skin and tissue assessment; preventive skin and tissue care; early mobilisation; use of pressure relief devices/support surfaces; health education. (Total number of people with a pressure injury prevention care plan)/(Total number of people at risk of pressure injuries) x100
Prevalence of pressure injuries | 15 months
  Number of patients presenting with a pressure injury at the start of care (Total number of people with one or more pressure injuries)/(Total number of people with health care provision) x100
Pressure injuries associated with care | 15 months
  Total number of people who develop one or more pressure injuries during care (Total number of people who develop one or more pressure injuries since admission or start of care)/(Total number of people with health care provision ) x 100
Healthcare-associated pressure injuries in persons at risk | 15 months
  Total number of persons who develop one or more pressure injuries during care and who had been assessed as being at risk of developing pressure injuries (Total number of persons developing one or more pressure injuries since admission or start of care)/(Total number of persons at risk of PBI with healthcare provision) x 100
Stage of most severe pressure injury: | 15 months
  Stage of the most severe pressure injury developed by patients classified as at risk or not at risk of developing pressure injuries.
Falls risk screening | 15 months
  Falls risk screening carried out on all patients aged 65 years and over to determine their risk of falling. (Total number of people with falls risk screening recorded)/(Total number of people) x100.
Multifactorial falls risk assessment | 15 months
  Multifactorial falls risk assessment carried out on patients at high risk of falls. This should include at least: mobility, activities of daily living and cognitive function (Total number of people with recorded falls risk assessment)/(Total number of people at risk of falls) x100.
Falls prevention care plan | 15 months
  Individualised falls and injury prevention plan for people at risk of falling, taking into account the scope of care and its possibilities, patient preferences and multifactorial assessment by professionals (Total number of people at high risk of falls with a recorded falls prevention care plan)/(Total number of people at high risk of falls) x100
Falls risk reassessment | 15 months
  Risk reassessments made after any significant change in health following a fall, at 30-90 days for people at high risk of falls or one year since the last reassessment for people at low risk. (Total number of people with falls risk reassessment recorded)/(Total number of people eligible for risk reassessment) x100
Exercise interventions | 15 months
  Considers whether people at risk of falls have been referred to a specialist for exercise or whether exercise interventions have been implemented. (Number of people at high risk of falls who have participated in @exercise and physical training interventions)/(Total number of people at high risk of falls where the indicator applies) x100
Number of falls | 15 months
  Number of falls that have occurred during the hospital stay or duration of care.(Total number of people who have fallen)/(Total number of people) x100
Injuries resulting from falls | 15 months
  Injuries resulting from the fall, according to the following scale: None, slight injury, moderate injury, severe injury, fear of falling, death. (Total number of persons with fall/s that have had consequences)/(Total number of persons who have fallen) x100
Urinary incontinence initial assessment | 15 months
  Initial assessment of presence of urinary incontinence. Total number of patients in whom the presence of urinary incontinence has been initially assessed, and who are registered / Total number of patients with positive detection of urinary incontinence during the data collection period) * 100
Voiding diary | 15 months
  Record of all urination and leakage for 3 consecutive days before and after the intervention. (Total number of patients with a voiding diary of 3 days recorded / Total number of patients with urinary incontinence discharged or attended during the data collection period) * 100
Scheduled urination | 15 months
  Using verbal and physical prompts or signals to make people pay attention to their dry/wet situation and the need to go to the bathroom. (Total number of patients with a scheduled urination care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Bladder training | 15 months
  Program of education and programmed evacuation in which the intervals of micturition are gradually adjusted. (Total number of patients with a bladder training care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Pelvic floor exercises | 15 months
  The individualized education and training of pelvic floor exercises. (Total number of patients with a pelvic floor exercise care plan, and it is registered / Total number of patients with urinary incontinence and a 3-day voiding diary discharged or attended in the data collection period) * 100
Severity | 15 months
  Severity of urinary incontinence. Total number of patients with different levels of urinary incontinence 24 hours prior to assessment / Total number of patients with urinary incontinence during the data collection period) x 100
Impact | 15 months
  Impact of urinary incontinence. (Total number of patients whose urinary incontinence has an impact on their quality of life, in the 24 hours prior to the assessment / Total number of patients with urinary incontinence during the data collection period) x 100
Improvement | 15 months
  Perception of improvement in urinary incontinence. (Total number of patients who perceive an improvement 6 weeks after the intervention / Total number of patients with urinary incontinence before the start of the intervention) x100
Comprehensive assessment (obesity) | 15 months
  Requires realization and documentation of a comprehensive assessment of children from birth to 12 years has been carried out considering all of the following elements: Growth; Feeding / breastfeeding (as appropriate); Physical activity; Sedentary behaviour / screen time; Family environment. (Number of children from birth to 12 years (and parents or carers) who have had a full assessment)/(Number of children from birth to 12 years ) x100.
Promotion of healthy behaviours | 15 months
  Delivery and documentation of age-appropriate healthy behaviour promotion recommendations (e.g.: Support for breastfeeding, exclusive or complementary feeding (if appropriate); Healthy behaviour promotion on feeding; Healthy behaviour promotion on physical activity; Healthy behaviour promotion on sedentary/ screen time. (Number of children from birth to 12 years (and parents/caregivers) who have received healthy behaviour promotion interventions)/(Number of children from birth to 12 years) x100
Education and support | 15 months
  Requires documented evidence that parents/primary caregivers have received age-appropriate education on any of the following topics: breastfeeding, role modelling, child feeding practices, family physical activity; screen time, physical activity, healthy eating. (Number of parents or caregivers of children from birth to 12 years who have been provided with education and support to maintain healthy habits)/(Number of children from birth to 12 years ) x100
Exclusive breastfeeding, children from birth to 6 months of age | 15 months
  Children from 0 to 183 days inclusive who have received exclusive breastfeeding, directly from the breast or stored. (Number of children 0-6 months (or-183 days) who received EXCLUSIVE breastfeeding in the previous 24 hours, and is registered / Total number of children 0-6 months with one or more visits well-infant-child follow-up in the previous year) x100
Breastfeeding, children from 6 months of age up to 2 years | 15 months
  Children with more than 183 days of life who received breastfeeding directly from the breast or stored. (Number of children >6 months and up to 2 years (more than 183 days-2 years) who received breastfeeding in the previous 24 hours, and is registered / Total number of children >6 months - and up 2 years with one or more well-infant-child follow-up visits in the previous year) x100
Daily physical activity | 15 months
  Number of children from birth from 0 to 12 years of age who meet the recommendations on amount of daily physical activity. (Number of children from birth to 12 years of age who meet the recommendations on amount of daily exercise, and are registered / Total number of children from birth to 12 years of age with one or more follow-up visits of the healthy infant-child in the previous year, with assessment of physical activity or comprehensive assessment) x100
Sedentary behaviour | 15 months
  Number of children from birth to 12 years old who spent the recommended time for their age in front of a screen. (Number of children from birth to 12 years old, whose daily screen time is the recommended for their age, as of parents' declaration, and is registered / Total number of children from births up to 12 years of age with one or more follow-up visits to the well-child infant in the previous year, with assessment of screen time or comprehensive assessment) x100
Fruit and vegetable intake | 15 months
  Number of children aged 2-12 consuming fruit and vegetables daily and up to 5 times a day, and recorded (Number of children aged 2-12 consuming fruit and vegetables daily or up to 5 times a day)/(Number of children aged 2-12 ) x100
Assessment of mother's intention to breastfeed | 15 months
  Requires that mothers of newborns have been assessed for their intention to breastfeed during hospital admission for delivery (Number of mothers assessed for their intention to breastfeed)/(Total number of mothers) x100
Postpartum assessment of breastfeeding | 15 months
  Assessment of breastfeeding completed within the first 24 hours of the newborn life. It should include all of the following components: knowledge and attitudes; level of self-efficacy or self-confidence regarding breastfeeding; concerns; support network; breastfeeding technique in relation to positioning, latch-on, effective milk transfer; assessment of the newborn/infant (regarding breastfeeding). To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed on the breastfeeding process in the first 24 hours/Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Skin-to-skin contact | 15 months
  Skin-to-skin contact is the placement of a newborn, naked or with a diaper and cap, in a prone position on the bare chest of a person, covered with a previously heated blanket to prevent heat loss. It should be facilitated immediately (up to 1 hour) after birth or once the child and the nursing person are clinically stable. (Number of infants performing skin-to-skin immediately after birth or with clinically stable dyad /Total number of infants) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Information and education on breastfeeding, and support for the breastfeeding process (hospital). | 15 months
  In Hospital Care, it is considered completed if postpartum training and resources have been provided to the mother by the interprofessional team on breastfeeding before hospital discharge. The specific components are: Latching/postpartum and latch-on; Milk transfer; Breastfeeding based on infant cues; Other. ((Number of mothers receiving information and education on breastfeeding and support for the breastfeeding process)/ Total number of dyads) x100 Dyad: Pair consisting of mother and breastfeeding infant who form a bond with each other.
Breastfeeding education and support for family members (hospital) | 15 months
  In hospital care, it is considered completed if education and support in breastfeeding has been carried out for family members before hospital discharge. (Number of dyads whose family has received education and support in breastfeeding / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Breastfeeding at first feeding | 15 months
  Requires the infant to have been breastfed for the first feeding after birth (Number of infants who were breastfed for the first feeding)/(Total number of infants discharged) x100
Type of breastfeeding of the newborn during the hospital stay | 15 months
  Type of breastfeeding of the newborn during the hospital stay. (Number of infants exclusively breastfed, receiving mixed breastfeeding or not breastfed during hospital stay / Total number of infants discharged) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Early assessment of breastfeeding in primary care | 15 months
  In Primary Care, early assessment is considered completed between hospital discharge and day 8 of the neonate's life (included). To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed early on the process of breastfeeding (between hospital discharge and 8 days of life / Total number of dyads between hospital discharge and 8 days of life of the newborn) x 100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Follow-up assessment of breastfeeding in primary care (from 9 days of life to 6 months) | 15 months
  In Primary Care, the follow-up evaluation is carried out between 9 days of life and 6 months/183 days of life of the neonate (included). To carry out the assessment, a breastfeeding assessment tool may be used. (Number of dyads assessed on the breastfeeding process from 9 days of life to 6 months / Total number of dyads from 9 days of life to 6 months of the newborn) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Breastfeeding education for the breastfeeding person (Primary care) | 15 months
  In Primary Care, it is considered completed if training has been carried out and resources have been provided to the mother after hospital discharge by the interprofessional team in breastfeeding, at least once in the period after discharge to 8 days or in the period from 9 days to 6 months, in the same visit or in successive visits. (Number of lactating persons receiving education in breastfeeding / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Breastfeeding education and support for family members | 15 months
  In Primary Care, it is considered accomplished if breastfeeding education and support has been provided to family members, at least once in the period after discharge to 8 days or in the period from 9 days to 6 months, in the same visit or on successive visits. (Number of dyads whose family has received education and support in breastfeeding / Total number of dyads) x100 Dyad: A couple formed by the mother and the nursing baby who form a bond with each other.
Type of breastfeeding of the newborn in early stage | 15 months
  Type of breastfeeding of the newborn from birth to 8 days of life assessed in Primary care. (Number of newborns who were exclusively breastfed, received mixed breastfeeding or were not breastfed from birth to 8 days of life / Total number of newborns between 0 and 8 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Type of breastfeeding of the newborn in follow-up 1 | 15 months
  Type of breastfeeding of the newborn from 9 to 90 days of life, assessed in Primary Care. (Number of infants exclusively breastfed, receiving mixed breastfeeding or not breastfed from 9 days to 90 days of life / Total number of infants from 9 to 90 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Type of breastfeeding of the newborn in follow-up 2 | 15 months
  Type of breastfeeding of the newborn from 91 to 182 days of life assessed in Primary care (Number of newborns who received exclusive breastfeeding, receiving mixed breastfeeding or not breastfed from 91 days to 182 days of life / Total number of newborns from 91 to 182 days of life) x100 Exclusive breastfeeding: The infant receives directly or indirectly breast milk. He does not receive any other type of solid or liquid food.
  Mixed breastfeeding: The infant receives breast milk as well as other solid and liquid foods (including water), including non-human milk or formula.
  Non-breastfeeding: The infant receives artificial milk and/or animal milk. The infant does not receive breast milk.
Exclusive breastfeeding at 6 months | 15 months
  Number of newborns who received exclusive breastfeeding on day 183 of life (Number of newborns who received exclusive breastfeeding on day 183 of life / Total number of newborns with 183 days completed) x100

SECONDARY OUTCOMES:
Type of institution | 15 months
  Hospital unit, primary care unit or nursing home unit.
Type of unit | 15 months
  Age, health problems and care required by the patients attended by the unit on a regular basis.
Team Leader rol | 15 monthts
  Supervisor, mid-level leader, high-level leader, clinical nurse, other rol in the institution
Team members rol | 15 months
  Supervisor, mid-level leader, high-level leader, clinical nurse, other rol in the institution
Date of discharge | 15 months
  Patients discharge date in case of hospital admissions.
Date of attention | 15 months
  Date when patients were attended in case of primary care.
Date of residence | 15 months
  Date when patients were a resident in case of socio-healthcare centres.
Patients Age | 15 months
  Age of patients.
Patients Sex | 15 months
  Sex of patients.
Type of incontinence | 15 months
  Type of incontinence presented by the patient who has been assessed as an incontinent patient. It may be stress, urge or mixed incontinence.
Incontinence triggering factors. | 15 months
  Factors that cause the patient to experience episodes of incontinence. They may be: Multifactorial causes (cognitive, previous urinary problems, neurological causes, malignancy, surgery); Medication; Overweight/Obesity; Tobacco use; Lifestyle and fluid intake.
Mother´s age | 15 months
  Age of the mother.
Breastfeeding for the first time | 15 months
  First time the mother is facing breastfeeding or not.
Type of birth | 15 months
  Way in which the newborn was born: vaginal delivery, instrumental birth, caesarean section.
Weeks of gestation | 15 months
  Number of weeks of pregnancy.
Weight at birth | 15 months
  Weight of the newborn at birth, measured in grams.
Child weight | 15 months
  Child's weight measured in kilograms.
Child's height | 15 months
  Child's height measured in centimetres.
Reason for admission/consultation | 15 months
  Reason for admission/consultation of patients. Reason for the patient to be admitted to the Hospital or to attend the consultation.
Previous history of pain | 15 months
  History of previous painful experiences of the patient.
Type of smoker | 15 months
  Currently smoking or have quit less than 1 month ago or non-active if quit more than 1 month ago but less than 6 months ago.
Smoking relapses | 15 months
  Number of relapses since patient stopped smoking
Previous of pressure injuries | 15 months
  Numbers of pressure injuries that the patient had at the start of care
Stage of change | 15 months
  Patient's stage of change according to Prochaska y Diclemente
Tobacco use | 15 months
  Number of cigarettes or derivatives consumed by the patient per day and year
Barriers | 15 months
  Barriers for the implementation of evidence-based recommendations in the units assessed using a questionnaire adapted from the The comprehensive, integrated checklist of determinants of practice (TICD checklist) and the Consolidated Framework for Implementation Research.
Strategies | 15 months
  Strategies designed for the implementation of evidence-based recommendations in the units assessed using a questionnaire adapted from the Expert Recommendations for Implementing Change (ERIC).
Evidence Based Practice competencies | 15 months
  Competencies in evidence-based practice of the healthcare professionals working in the units that are implementing evidence-based recommendations, assessed with the questionnaire EBP-COQ Prof©.
Clinical leadership skills | 15 months
  Clinical leadership skills of the healthcare professionals working in the units that are implementing evidence-based recommendations, assessed with the clinical leadership survey©.
Empowerment | 15 months
  Empowerment of the healthcare professionals working in the units that are implementing evidence-based recommendations, assessed with the Conditions for Work Effectiveness Questionnaire - II ©.
Evidence Based Practice (EBP) climate and leadership | 15 months
  EBP climate and leadership in the units participating in the project measured with the evidence-based practice nursing leadership and work environment scales ©.
Professional's sex | 15 months
  Sex of the professionals participating in the local implementation team
Professional's age | 15 months
  Age of the professionals participating in the local implementation team
Professional's qualifications | 15 months
  Professional's qualifications of the professionals participating in the local implementation team
Professional's experience | 15 months
  Professional's experience of the professionals participating in the local implementation team

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Moreno-Casbas, PhD, Study Director — Instituto de Salud Carlos III; Esther González-María, PhD, Principal Investigator — Instituto de Salud Carlos III; Leticia Bernués-Caudillo, PhD Candidate, Study Chair — Instituto de Salud Carlos III; Laura Albornos-Muñoz, PhD, Study Chair — Instituto de Salud Carlos III; Alba Ayala, PhD, Study Chair — Instituto de Salud Carlos III
Locations (1):
- Instituto de Salud Carlos III - Unidad de Investigación en Cuidados y Servicios de Salud, Madrid, Spain

REFERENCES:
- [Background] Kreindler SA. What if implementation is not the problem? Exploring the missing links between knowledge and action. Int J Health Plann Manage. 2016 Apr;31(2):208-26. doi: 10.1002/hpm.2277. Epub 2014 Nov 25. PMID 25424863
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Squires JE, Estabrooks CA, Gustavsson P, Wallin L. Individual determinants of research utilization by nurses: a systematic review update. Implement Sci. 2011 Jan 5;6:1. doi: 10.1186/1748-5908-6-1. PMID 21208425
- [Background] Meijers JM, Janssen MA, Cummings GG, Wallin L, Estabrooks CA, Y G Halfens R. Assessing the relationships between contextual factors and research utilization in nursing: systematic literature review. J Adv Nurs. 2006 Sep;55(5):622-35. doi: 10.1111/j.1365-2648.2006.03954.x. PMID 16907795
- [Background] Ortuno-Soriano I, Munoz-Jimenez D, Moreno-Casbas T, Albornos-Munoz L, Gonzalez-Maria E; en nombre del Grupo de Trabajo del Programa de implantacion de buenas practicas en Centros Comprometidos con la Excelencia en Cuidados(R). Evaluation of implementation strategies of the Best Practices Spotlight Organisations (BPSO) Project in Spain. Enferm Clin (Engl Ed). 2020 May-Jun;30(3):222-230. doi: 10.1016/j.enfcli.2019.10.027. Epub 2020 May 7. English, Spanish. PMID 32389600
- [Background] Powell BJ, Fernandez ME, Williams NJ, Aarons GA, Beidas RS, Lewis CC, McHugh SM, Weiner BJ. Enhancing the Impact of Implementation Strategies in Healthcare: A Research Agenda. Front Public Health. 2019 Jan 22;7:3. doi: 10.3389/fpubh.2019.00003. eCollection 2019. PMID 30723713
- [Background] Lewis CC, Boyd MR, Walsh-Bailey C, Lyon AR, Beidas R, Mittman B, Aarons GA, Weiner BJ, Chambers DA. A systematic review of empirical studies examining mechanisms of implementation in health. Implement Sci. 2020 Apr 16;15(1):21. doi: 10.1186/s13012-020-00983-3. PMID 32299461
- [Background] Allen P, Pilar M, Walsh-Bailey C, Hooley C, Mazzucca S, Lewis CC, Mettert KD, Dorsey CN, Purtle J, Kepper MM, Baumann AA, Brownson RC. Quantitative measures of health policy implementation determinants and outcomes: a systematic review. Implement Sci. 2020 Jun 19;15(1):47. doi: 10.1186/s13012-020-01007-w. PMID 32560661
- [Background] Moreno-Casbas T. Perspectives: Implementation strategies to adopt and integrate evidence-based nursing. What are we doing? J. Res. Nurs. 2015;20:729-33.
- [Background] Lau R, Stevenson F, Ong BN, Dziedzic K, Treweek S, Eldridge S, Everitt H, Kennedy A, Qureshi N, Rogers A, Peacock R, Murray E. Achieving change in primary care--causes of the evidence to practice gap: systematic reviews of reviews. Implement Sci. 2016 Mar 22;11:40. doi: 10.1186/s13012-016-0396-4. PMID 27001107
- [Background] Almazrou SH, Alfaifi SI, Alfaifi SH, Hakami LE, Al-Aqeel SA. Barriers to and Facilitators of Adherence to Clinical Practice Guidelines in the Middle East and North Africa Region: A Systematic Review. Healthcare (Basel). 2020 Dec 15;8(4):564. doi: 10.3390/healthcare8040564. PMID 33333843
- [Background] Davies B, Edwards N, Ploeg J, Virani T. Insights about the process and impact of implementing nursing guidelines on delivery of care in hospitals and community settings. BMC Health Serv Res. 2008 Feb 2;8:29. doi: 10.1186/1472-6963-8-29. PMID 18241349
- [Background] Ploeg J, Davies B, Edwards N, Gifford W, Miller PE. Factors influencing best-practice guideline implementation: lessons learned from administrators, nursing staff, and project leaders. Worldviews Evid Based Nurs. 2007;4(4):210-9. doi: 10.1111/j.1741-6787.2007.00106.x. PMID 18076464
- [Background] Mickan S, Burls A, Glasziou P. Patterns of 'leakage' in the utilisation of clinical guidelines: a systematic review. Postgrad Med J. 2011 Oct;87(1032):670-9. doi: 10.1136/pgmj.2010.116012. Epub 2011 Jun 29. PMID 21715571
- [Background] Fleiszer AR, Semenic SE, Ritchie JA, Richer MC, Denis JL. A unit-level perspective on the long-term sustainability of a nursing best practice guidelines program: An embedded multiple case study. Int J Nurs Stud. 2016 Jan;53:204-18. doi: 10.1016/j.ijnurstu.2015.09.004. Epub 2015 Sep 8. PMID 26453418
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N. Tailored interventions to overcome identified barriers to change: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005470. doi: 10.1002/14651858.CD005470.pub2. PMID 20238340
- [Background] Flodgren G, Deane K, Dickinson HO, Kirk S, Alberti H, Beyer FR, Brown JG, Penney TL, Summerbell CD, Eccles MP. Interventions to change the behaviour of health professionals and the organisation of care to promote weight reduction in overweight and obese people. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD000984. doi: 10.1002/14651858.CD000984.pub2. PMID 20238311
- [Background] Esposito P, Dal Canton A. Clinical audit, a valuable tool to improve quality of care: General methodology and applications in nephrology. World J Nephrol. 2014 Nov 6;3(4):249-55. doi: 10.5527/wjn.v3.i4.249. PMID 25374819
- [Background] Wentland BA, Hinderer KA. A Nursing Research and Evidence-Based Practice Fellowship Program in a Magnet(R)-designated pediatric medical center. Appl Nurs Res. 2020 Oct;55:151287. doi: 10.1016/j.apnr.2020.151287. Epub 2020 May 15. PMID 32482374
- [Background] Holmes BJ, Best A, Davies H, Hunter D, Kelly MP, Marshall M, Rycroft-Malone J. Mobilising knowledge in complex health systems: A call to action. Evid. Policy 2017;13:539-60.
- [Background] Powell BJ, McMillen JC, Proctor EK, Carpenter CR, Griffey RT, Bunger AC, Glass JE, York JL. A compilation of strategies for implementing clinical innovations in health and mental health. Med Care Res Rev. 2012 Apr;69(2):123-57. doi: 10.1177/1077558711430690. Epub 2011 Dec 26. PMID 22203646
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Sinuff T, Muscedere J, Rozmovits L, Dale CM, Scales DC. A qualitative study of the variable effects of audit and feedback in the ICU. BMJ Qual Saf. 2015 Jun;24(6):393-9. doi: 10.1136/bmjqs-2015-003978. Epub 2015 Apr 27. PMID 25918432
- [Background] Munoz Jimenez D. From evidence-based nursing to healthcare practice: The evaluation of results as an integrating element. Enferm Clin (Engl Ed). 2018 May-Jun;28(3):149-153. doi: 10.1016/j.enfcli.2018.04.004. No abstract available. English, Spanish. PMID 29778244
- [Background] Christina V, Baldwin K, Biron A, Emed J, Lepage K. Factors influencing the effectiveness of audit and feedback: nurses' perceptions. J Nurs Manag. 2016 Nov;24(8):1080-1087. doi: 10.1111/jonm.12409. Epub 2016 Jun 16. PMID 27306646
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Duenas M, Salazar A, Ojeda B, Fernandez-Palacin F, Mico JA, Torres LM, Failde I. A nationwide study of chronic pain prevalence in the general spanish population: identifying clinical subgroups through cluster analysis. Pain Med. 2015 Apr;16(4):811-22. doi: 10.1111/pme.12640. Epub 2014 Dec 19. PMID 25530229
- [Background] García FJ, Salinas J, Madurga B, Cózar JM, Esteban M. Guía de atención a personas con incontinencia urinaria [internet]. Madrid: Asociación Española de Urología; Enero 2020 [consultado abril de 2021]. Available in: https://www.consejogeneralenfermeria.org/documentos-de-interes/guias-clinicas/send/67-guias-clinicas/908-guia-de-atencion-a-personas-con-incontinencia-urinaria
- [Background] Dufour S, Wu M. No. 397 - Conservative Care of Urinary Incontinence in Women. J Obstet Gynaecol Can. 2020 Apr;42(4):510-522. doi: 10.1016/j.jogc.2019.04.009. PMID 32303295
- [Background] Estudio ALADINO 2019: Estudio sobre Alimentación, Actividad Física, Desarrollo Infantil y Obesidad en España 2019. Agencia Española de Seguridad Alimentaria y Nutrición. Ministerio de Consumo. Madrid, 2020
- [Background] Departamento de Salud del Gobierno Vasco. Estrategia de prevención de la obesidad infantil en Euskadi. PLAN SANO. 2019. Editado por Servicio Central de publicaciones del Gobierno Vasco. Disponible en: https://www.euskadi.eus/estrategia/prevencion-de-la-obesidad-infantil-en-euskadi/web01-a2osabiz/es/
- [Background] World Health Organization. Infant and young child feeding. Ginebra: WHO; 2021 [acceso12/11/2021]. Disponible en: https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding.
- [Background] Encuesta Nacional de Salud de España 2017. Instituto nacional de estadística. [acceso 25/08/2019]. Available in: https://www.mscbs.gob.es/estadEstudios/estadisticas/encuestaNacional/encuesta2017.htm
- [Background] OMS, Ministerio de Sanidad. La higiene de las manos en la asistencia ambulatoria y domiciliaria y en los cuidados de larga duración. Guía de aplicación de la estrategia multimodal de la OMS para la mejora de la higiene de las manos y del modelo
- [Background] Agencia Española del Medicamento y Producto Sanitarios. Programa Higiene de manos del SNS. Informe de indicadores 2019. Madrid. 2020
- [Background] Estudio nacional de vigilancia de infección nosocomial en servicios de medicina intensiva. Vall d'hebron. Barcelona; 2019. Available in: https://hws.vhebron.net/envin-helics/
- [Background] Estudio APEAS. Estudio sobre la seguridad de los pacientes en atención primaria de salud. Madrid: Ministerio de Sanidad y Consumo; 2008.
- [Background] Flottorp SA, Oxman AD, Krause J, Musila NR, Wensing M, Godycki-Cwirko M, Baker R, Eccles MP. A checklist for identifying determinants of practice: a systematic review and synthesis of frameworks and taxonomies of factors that prevent or enable improvements in healthcare professional practice. Implement Sci. 2013 Mar 23;8:35. doi: 10.1186/1748-5908-8-35. PMID 23522377
- [Background] Escobar-Aguilar G, Moreno-Casbas MT, Gonzalez-Maria E, Martinez-Gimeno ML, Sanchez-Pablo C, Orts-Cortes I. The SUMAMOS EXCELENCIA Project. J Adv Nurs. 2019 Jul;75(7):1575-1584. doi: 10.1111/jan.13988. Epub 2019 Apr 2. PMID 30816569
- [Background] Martinez-Gimeno ML, Fernandez-Martinez N, Escobar-Aguilar G, Moreno-Casbas MT, Brito-Brito PR, Caperos JM. SUMAMOS EXCELENCIA(R) Project: Results of the Implementation of Best Practice in a Spanish National Health System (NHS). Healthcare (Basel). 2021 Mar 28;9(4):374. doi: 10.3390/healthcare9040374. PMID 33800670
- [Background] Ministerio de Sanidad - Gobierno de España. Encuesta sobre alcohol y otras drogas en ESpaña (EDADES) 1995-2022. 2022.
- [Background] Ministerio de Sanidad - Gobierno de España. Muertes atribuibles al consumo de tabaco en España, 2000-2014. 2017.
- [Background] VH R, LF S. Intervenciones de enfermería para el abandono del hábito de fumar (Cochrane). La Bibl Cochrane Plus. 2008;2.
- [Background] Lindson N, Pritchard G, Hong B, Fanshawe TR, Pipe A, Papadakis S. Strategies to improve smoking cessation rates in primary care. Cochrane Database Syst Rev. 2021 Sep 6;9(9):CD011556. doi: 10.1002/14651858.CD011556.pub2. PMID 34693994
- [Background] Pancorbo-Hidalgo PL, García-Fernández FP, Pérez-López C y Soldevilla Agreda JJ. Prevalencia de lesiones por presión y otras lesiones cutáneas relacionadas con la dependencia en población adulta en hospitales españoles: resultados del 5º Estudio Nacional de 2017. Available in: https://gneaupp.info/wp-content/uploads/2021/11/30-2-2019-076.pdf
- [Background] García-Fernández F.P, Torra i Bou J.E, Soldevilla-Agreda JJ, Verdú Soriano J, Torra i Bou J.E. Prevalencia de lesiones por presión y otras lesiones cutáneas relacionadas con la dependencia en centros de atención primaria de salud de España en 2017. Available in: http://gerokomos.com/wp-content/uploads/2019/10/30-3-2019-134.pdf
- [Background] Soldevilla-Agreda JJ, García-Fernández F.P, Rodríguez-Palma M, Pancorbo Hidalgo PL. Prevalencia de lesiones por presión y otras lesiones cutáneas relacionadas con la dependencia en residencias de mayores y centros sociosanitarios de España en 2017. Gerokomos. 2019;30(4):192-199. Available in: http://gerokomos.com/wp-content/uploads/2019/12/30-4-2019-192.pdf
- [Background] Estrategia de Seguridad del Paciente del Sistema Nacional de Salud Período 2015-2020. Comité Institucional de la Estrategia de Seguridad del Paciente. Consejo Interterritorial del Sistema Nacional de Salud del día 29 de julio de 2015. Ministerio de Sanidad, Servicios Sociales e Igualdad. Available in: https://seguridaddelpaciente.sanidad.gob.es/docs/Estrategia_Seguridad_del_Paciente_2015-2020.pdf
- [Background] Sinn CL, Tran J, Pauley T, Hirdes J. Predicting Adverse Outcomes After Discharge From Complex Continuing Care Hospital Settings to the Community. Prof Case Manag. 2016 May-Jun;21(3):127-36; quiz E3-4. doi: 10.1097/NCM.0000000000000148. PMID 27035083
- [Background] Pancorbo-Hidalgo, P. L., García-Fernández, F. P., Torra i Bou, J.-E., Verdú Soriano, J., & Soldevilla-Agreda, J. J. (2014). Epidemiología de las úlceras por presión en España en 2013: 4.o Estudio Nacional de Prevalencia. Gerokomos, 25(4), 162-170.
- [Background] Jiang Q, Li X, Qu X, Liu Y, Zhang L, Su C, Guo X, Chen Y, Zhu Y, Jia J, Bo S, Liu L, Zhang R, Xu L, Wu L, Wang H, Wang J. The incidence, risk factors and characteristics of pressure ulcers in hospitalized patients in China. Int J Clin Exp Pathol. 2014 Apr 15;7(5):2587-94. eCollection 2014. PMID 24966973
- [Background] Rubenstein LZ, Josephson KR. The epidemiology of falls and syncope. Clin Geriatr Med. 2002 May;18(2):141-58. doi: 10.1016/s0749-0690(02)00002-2. PMID 12180240
- [Background] World Health Organization. WHO global report on falls prevention in older age. 2007. Available in: https://www.who.int/publications/i/item/9789241563536
- [Background] Rubenstein LZ, Powers CM, MacLean CH. Quality indicators for the management and prevention of falls and mobility problems in vulnerable elders. Ann Intern Med. 2001 Oct 16;135(8 Pt 2):686-93. doi: 10.7326/0003-4819-135-8_part_2-200110161-00007. No abstract available. PMID 11601951
- [Background] LeLaurin JH, Shorr RI. Preventing Falls in Hospitalized Patients: State of the Science. Clin Geriatr Med. 2019 May;35(2):273-283. doi: 10.1016/j.cger.2019.01.007. Epub 2019 Mar 1. PMID 30929888
- See also: Project website — https://evidenciaencuidados.isciii.es/sumamos-excelencia-2024-2025/